CLINICAL TRIAL: NCT06952842
Title: A Single-Arm, Open-Label, Phase 1/2 Clinical Trial of ZVS203e in Subjects With Retinitis Pigmentosa Associated With RHO Mutation
Brief Title: Safety and Efficacy of ZVS203e in the Treatment of Retinitis Pigmentosa Caused by RHO Gene Mutation
Acronym: ZVS203e
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chigenovo Co., Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYB-2025-001
Record Dates: First submitted 2025-04-22; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Retinitis Pigmentosa
Keywords: Gene editing; ZVS203e; RHO; Retinitis pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): All patients enrolled in the study will receive a single subretinal injection of ZVS203e in one eye
  Interventions: Drug: ZVS203e

INTERVENTIONS:
Drug: ZVS203e — ZVS203e injection is a clear, transparent liquid containing a recombinant adeno-associated virus serotype 8 (rAAV8) vector that expresses humanized SauriCas9 protein and single guide RNA (sgRNA) targeting specific mutations in the RHO gene.
  Other Names: rAAV8

SUMMARY:
This trial employs a single-arm, open-label seamless Phase I/II design, consisting of two stages: Phase I dose exploration and Phase II dose expansion.The primary objective of this trial is to evaluate the safety, tolerability, and efficacy of subretinal injection of ZVS203e solution.

DETAILED DESCRIPTION:
ZVS203e injection is administered via a single subretinal injection of rAAV8 vector carrying CRISPR/Cas9 gene-editing tools to silence mutated genes, allowing retinal cells to express only normal functional proteins, thereby treating RHO-adRP.

This trial employs a single-arm, open-label seamless Phase I/II design, consisting of two stages: Phase I dose escalation and Phase II dose expansion, with an anticipated total enrollment of 9 to 18 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical diagnosis of retinitis pigmentosa (RP) (aged 18 years or older);
2. RHO (c.403C>T, p.R135W) gene site-specific mutation was confirmed by genetic testing, and no other ophthalmic genetic diseases were complicated;
3. The researchers judged that the target eye had viable retinal photoreceptor cells and retinal pigment epithelial cells;
4. The best corrected visual acuity of the target eye is between 2.0 LogMAR and 0.5 LogMAR (including 2.0 LogMAR and 0.5 LogMAR, which is equivalent to a number of fingers to 60 letters);
5. The subject and his or her spouse agree to use effective contraception during the trial period and for at least 1 year after dosing;
6. Voluntarily participate in clinical trials and sign informed consent, and can complete the whole test process according to the protocol requirements.

Exclusion Criteria:

1. The researcher determined that the target eye currently has or had macular lesions such as macular hiatal hole or macular neovascularization;
2. Have other eye conditions that may prevent surgery or interfere with interpretation of the study endpoint, such as glaucoma, diabetic retinopathy, eye or periocular infections, active endophthalmitis, etc.
3. Within 3 months prior to enrollment, the study eye had received any intraocular surgery, such as phacoemulsification cataract extraction.
4. The study eye had undergone retinal reattachment or vitrectomy.
5. Participants who had participated in any drug or medical device clinical trial within 3 months before enrollment;
6. Previously treatment of either eye with gene therapy or stem cell therapy for RP and other ocular diseases, including but not limited to viral vector gene therapy, RNA therapy.
7. Treatment with medications that may affect the efficacy and safety evaluation of the investigational product within 3 months prior to enrollment (e.g., ranibizumab, bevacizumab, aflibercept, conbercept).
8. Known allergy to the drug planned to be used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-18 (Estimated); Primary Completion 2030-06-18 (Estimated); Study Completion 2045-06-18 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of subretinal injection of ZVS203e solution | 24 weeks post-treatment
  Types, severity, and incidence of adverse events (AE) and serious adverse events (SAE) in the eyes and throughout the body within 24 weeks post-treatment, including dose-limiting toxicities (DLT) during the dose escalation phase.
Change from baseline in best-corrected visual acuity (BCVA) | 24 weeks post-treatment
  Change in best-corrected visual acuity (BCVA) of the treated eye at 24 weeks compared to baseline.

SECONDARY OUTCOMES:
Change from Baseline in Visual function metrics | 24 weeks post-treatment
  Treatment outcomes for visual function metrics include changes from baseline in LLVA, dynamic visual field, microperimetry, FST, contrast sensitivity, color vision, and mfERG; as well as changes from baseline in the NEI-VFQ-25 score reported by the participants.
Change from Baseline in OCT | 24 weeks post-treatment
  Compare changes in retinal morphology and alterations in cell layers of the retina before and after drug administration.
Evaluate the immunogenicity of ZVS203e | 24 weeks post-treatment
  Changes in SauriCas9 antibody, AAV8 antibody, and neutralizing antibody levels from baseline in the subjects.
Evaluate the pharmacokinetic characteristics of ZVS203e | 24 weeks post-treatment
  Changes in AAV8 vector DNA and mRNA levels in the blood and tears of participants compared to baseline.
Change from Baseline in multi-luminance mobility test (MLMT) | 24 weeks post-treatment
  MLMT was assessed using both eyes at 1 or more of 7 levels of illumination, ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night).

CONTACTS AND LOCATIONS:
Overall Officials: Hongliang Dou, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu X, Jia R, Meng X, Li Y, Yang L. Retinal degeneration in humanized mice expressing mutant rhodopsin under the control of the endogenous murine promoter. Exp Eye Res. 2022 Feb;215:108893. doi: 10.1016/j.exer.2021.108893. Epub 2021 Dec 14. PMID 34919893
- [Background] Liu X, Qiao J, Jia R, Zhang F, Meng X, Li Y, Yang L. Allele-specific gene-editing approach for vision loss restoration in RHO-associated retinitis pigmentosa. Elife. 2023 Jun 5;12:e84065. doi: 10.7554/eLife.84065. PMID 37272616